CLINICAL TRIAL: NCT06141187
Title: Percutaneous Vertebroplasty Vs. Sham for Osteoporotic Vertebral Compression Fractures Focusing on Pain and Economy: a Single-center, Double-blind Randomized Controlled Clinical Trial
Brief Title: Percutaneous Vertebroplasty Vs. Sham for Osteoporotic Vertebral Compression Fractures Focusing on Pain and Economy.
Acronym: VOPE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS/KIR 012/2023
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-04

CONDITIONS: Osteoporotic Fractures; Vertebral Fracture
Keywords: vertebroplasty; Pain
MeSH Terms: conditions — Osteoporotic Fractures; Spinal Fractures; Pain | interventions — Vertebroplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vertebroplasty (Active Comparator): Polymethyl-methacrylate (PMMA) cement is prepared and injected slowly into the vertebral body under constant bi-plane fluoroscopy
  Interventions: Procedure: Vertebroplasty
- Sham vertebroplasty (Sham Comparator): A short needle is passed through the skin, but not as far as the periosteum. PMMA is mixed to mimic the PVP procedure but not injected into the vertebral body.
  Interventions: Procedure: Sham Vertebroplasty

INTERVENTIONS:
Procedure: Vertebroplasty — PVP
  Arms: Vertebroplasty
Procedure: Sham Vertebroplasty — Sham PVP
  Arms: Sham vertebroplasty

SUMMARY:
The purpose of this randomized double-blind clinical trial is to determine the efficacy of percutaneous vertebroplasty (PVP) in relieving severe pain in patients with MRI-verified acute or sub-acute osteoporotic vertebral compression fractures (OVCFs) compared to sham as well as examine the socio-economic implications associated with performing vertebroplasty.

The primary outcome is improvement of pain intensity as measured on a Visual Analog Scale (VAS, 0 to100) 12 weeks after treatment. Secondary outcomes include patient-reported back-related disability, patient-reported quality of life, spinal sagittal balance, complications associated with the procedure, incidence of new OVCFs and socioeconomic costs.

DETAILED DESCRIPTION:
The study design is a prospective, double-blind, randomized, sham-controlled clinical trial where patients are stratified into either involvement of 1-2 vertebral levels or 3-4 levels and randomized to either vertebroplasty or a sham operation. The trial is designed in accordance with the SPIRIT guidelines.

Patients will be examined in the outpatient clinic at the Center for Spine Surgery and Research, Lillebaelt Hospital, Kolding, Denmark. MRI scans and X-ray images will be performed at the radiology department at the hospital. Experienced neuro-radiologists carry out image analyses.

Spine surgeons who are experienced in PVP will perform the surgical procedures. Anaesthesiologists and spine surgeons are present at the facility in case of complications, following recommendations by the National Health Authority and have the capacity/capability to decompress the spinal canal in case of cement leakage.

Study subjects will be recruited from patients diagnosed with painful x-ray verified vertebral compression fractures in the Region of southern Denmark. The patients will be identified and referred to the trial site by the patients' general practitioner, chiropractor, physiotherapist, or from hospital inpatient and emergency departments in the region of Southern Denmark.

Subjects will initially be stratified into two groups based on the number of OVCFs into 1-2 levels or 3-4 levels. Within each of these two groups, randomization sheets in varying blocks of 8 with an equal number of PVP and sham patients in each block will be generated using software (www.randomizer.org) and will be placed in numbered, opaque, sealed envelopes. Treatment group assignment will be performed by a scrub nurse in the surgical theatre after the patient is draped but prior to skin incision. Throughout the trial, only the surgeon and the OR-nurse will have knowledge of the treatment assignment. The patient and all assessors remain blinded to the treatment group throughout the study.

During hospitalization, perioperative data on operation time, theater time and complications will be collected from the operating room staff during surgery. Upon discharge, length of stay will be recorded for each patient. After discharge, all visits to the outpatient clinic, either to the surgeon, nurse or physiotherapist as well as phone calls with questions regarding their procedure to the surgical nurse and time spent will be recorded.

Patients will be seen in the clinic for evaluation at 4, 12, and 52 weeks after treatment. MRI and full-standing anteroposterior and lateral radiographs will be taken at the 12-week follow-up time point. This will allow for identification of any healing at the index level as well as any new-onset OVCFs.

Treatment effectiveness analyses of the randomized trial data will performed on an intent-to-treat basis. Enrolled patients and outcome assessors will remain blinded for the duration of the trial. The 12-week follow-up will be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50+ and diagnosed with symptomatic osteoporotic spinal compression fractures between T6 and L5 (incl).
* Focal tenderness on the level of the vertebral fracture.
* Fractures verified with oedema of the relevant vertebra on the MRI STIR sequence
* Osteoporotic Fractures type 1-4.
* Fracture involves no more than 4 vertebral body levels.
* PVP can be done in one session.
* Back pain score measured on a Visual Analog Scale (VAS, 0 to 100) ≥ 60.
* Able to understand and read Danish.
* Written informed consent.
* Relevant pain started ≤ 3 months prior to enrollment.

Exclusion Criteria:

* - Contra-indications for spine surgery.
* Platelets < 30 mia/l.
* Osteoporotic Fractures type 5 and Pincer-type.
* Complete collapse of the vertebral body precluding insertion of needle.
* Presence of neurologic deficit.
* Contraindications for MRI scanning.
* Psychological or psychiatric disorder that is expected to interfere with compliance.
* Active malignancy.
* Mini Mental State Examination (MMSE) test score below 24.
* History of chronic back pain requiring ongoing opiate use.
* Systemic or local infection of the spine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity using the 100-point VAS | VAS will be recorded at time of randomization and after 1, 2, 3, 4 and 5 days, and after 2, 4, 8 and 12 weeks, and finally at 12 months and 24 months post-randomization
  Self-reported average pain intensity over the previous 24 hours, using the 100-point VAS will be recorded at time of randomization and after 1, 2, 3, 4 and 5 days, and after 2, 4, 8 and 12 weeks, and finally at 12 months and 24 months post-randomization

SECONDARY OUTCOMES:
Patient-reported disability. | Recorded at enrolment and at 4 and 12 weeks, 12 and 24 months post-randomization
  The patients rate their disability at the time of enrolment and at 4 and 12 weeks, 12 and 24 months post-randomization using the Oswestry Disability Index (ODI) questionnaire
Health-related quality of life. | Recorded at enrolment and at 4 and 12 weeks, 12 and 24 months post-randomization
  HRQL on the EuroQol 5-dimension 5-level (EQ-5D-5L)
Global Perceived Effect scale | Recorded at 4 and 12 weeks, 12 and 24 months post-randomization
  Global perceived effect of the treatment will be assessed using single question with seven-point descriptive scaling with the answers
Sagittal balance | Recorded at enrolment and 12 months post-randomization
  Full-length 36" lateral scoliosis radiographs taken with hands placed on the clavicles will be obtained to measure Pelvic Incidence, Pelvic Tilt, Sacral Slope, C7-Plumb Line and Lumbar Lordosis/Thoracic Kyphosis both preoperatively and after 12 months
Societal costs of treatment | Recorded 1 day at discharge and 12 months post-randomization
  The intervention costs will be obtained using data from hospital registries about outpatient contacts, inpatient admissions and length of stay, staff time for surgical procedure, recovery and rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Ø Andersen, MD, Principal Investigator — Sygehus Lillebælt
Locations (1):
- Rygcenter Syddanmark, Middelfart, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No
When the project is terminated, data from the project database will be archived at the Danish National Archives, and the research group will save an anonymized version of patient information from the database. After the project results are published, interested researchers will have two options for re-use of the data: upon receiving required permits they may apply for data extracts from DaneSpine and from the Danish National Archives - or they may receive anonymized raw data from DaneSpine and the project data base from us

REFERENCES:
- [Derived] Andersen MO, Andresen AK, Hartvigsen J, Hermann AP, Sorensen J, Carreon LY. Vertebroplasty for painful osteoporotic vertebral compression fractures: a protocol for a single-center doubled-blind randomized sham-controlled clinical trial. VOPE2. J Orthop Surg Res. 2024 Nov 30;19(1):813. doi: 10.1186/s13018-024-05301-x. PMID 39614265